CLINICAL TRIAL: NCT05261477
Title: Brain Injury Education and Outpatient Navigation for Hispanic Children and Their Caregivers-1stBIEN
Brief Title: Brain Injury Education and Outpatient Navigation-1stBIEN
Acronym: 1st-BIEN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Seattle Children's Hospital (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Nathalia Jimenez MD, MPH, Associate Professor Anesthesiology and Pain Medicine, Seattle Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: STUDY00003331; R01HD103700-01A1 (NIH)
Record Dates: First submitted 2022-01-24; First posted 2022-03-02 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Brain Injuries, Traumatic; Rehabilitation
Keywords: Hispanic or Latino; Child; Brain Injuries, Traumatic; Patient Navigation; Rehabilitation
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Intervention Model Description: Intervention group will receive one in-person education session, bi-weekly video reviews tailored to the child's injury and therapies; and, 3 months of bilingual outpatient navigation, using three way calls to model and coach problem solving skills, with parents as active participants. Attention control group will receive one in person-education session, monthly non-TBI (Well-child) texts and usual institutional follow up care. Participants in the control group do not receive video education or patient navigation.
Who Masked: Outcomes Assessor
Masking Description: All families enrolled in the trial will receive follow-up telephone assessments at 3-, 6-, and 12-months after discharge from the hospital. Follow-up interviews will be conducted by research assistants from the Social Development Research Group, who will be blinded to participant's study group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Intervention group receives one in person education session using the 1stBIEN booklet, video education via mobile phones and care coordination from a bilingual Patient Navigator-PN for 3-months. PN follow up patients weekly for the first month and once a month for two months. Video education is done weekly. Videos cover problem solving training, brain injury concepts, rehabilitation treatments and school resources individualized to patient and family needs. PNs facilitate transition to outpatient care, follow-up with specialists and primary care providers; use of community resources; and communication with teachers and school administrators. PN provides observational and experiential learning opportunities for parents, using three way calls for scheduling of services and interactions with clinics and schools. PN calls use a problem-solving training format, to reinforce parental experiential learning and improve self-efficacy. Expert MD providers (Co-investigators) will supervise PNs.
  Interventions: Behavioral: Bilingual Brain Injury Education and outpatient Navigation for Hispanic families
- Attention Control group (No Intervention): Attention Control group receives one in person education session using the 1stBIEN booklet, monthly well-child texts and usual post-injury care including routine follow-up by specialists and primary care providers, per guidelines at each recruiting institution. Control patients have access to a list of community resources included in the 1stBIEN booklet. While education using the 1stBIEN booklet is not part of the current usual care at participating institutions, providing all families with initial education at the time of discharge addresses ethical and practical considerations. It standardizes discharge processes at participating institutions while delineating differences in the intensity of education and care coordination activities.

INTERVENTIONS:
Behavioral: Bilingual Brain Injury Education and outpatient Navigation for Hispanic families — 1st BIEN was informed by Hispanic parents and clinical providers working with them. It considers their specific needs including lack of familiarity with shared decision models and of knowledge about patient rights and eligibility for community and school services. Based on principles of Social Cognitive Theory, 1st BIEN provides TBI education, teaches problem-solving skills to promote self-efficacy and advocacy; and provides outpatient navigation that allows for observational and experiential learning while supporting access to services in a timely manner. Central to the development of our intervention is the recognition of heterogeneity in individuals' level of readiness to adopt a health behavior according to their level of self-efficacy, expectations, and environment. The 1stBIEN intervention flexibly reduces barriers to access care, and simultaneously improves parental knowledge, health literacy, and self-efficacy to optimize outcomes.
  Other Names: 1stBIEN
  Arms: Intervention group

SUMMARY:
Traumatic brain injury (TBI) is a significant problem for U.S. Hispanic children. Compared to non-Hispanic children, Hispanic children have higher long-term disability and lower health related quality of life, even though differences are not present at hospital discharge. Rehabilitation decreases disability, but needs timely initiation, and long treatments in hospitals, community healthcare facilities and schools. Parents play a key role in their child's recovery. Hispanic parents face additional barriers to initiate and maintain outpatient treatments. They report knowledge gaps in TBI-education, community, and school support systems; language and health literacy barriers. The investigators developed, a bilingual bicultural theory-based program for Hispanic families consisting of Brain Injury Education and outpatient care Navigation (1st BIEN). It integrates in-person education enriched by video content delivered through mobile phones, with navigation during transitions to outpatient care and school return. The pilot established feasibility and acceptability of the program. This randomized control trial will determine efficacy to maintain long-term adherence to rehabilitation and reduce disability. It will enroll 150 parent-child dyads: children (6-17 y), with mild-complicated, moderate-severe TBI in 5 centers in Washington, Texas, Dallas, Utah and Oregon and their parents. Intervention group parents receive: One in-person education session, plus bi-weekly videos tailored to the child's TBI and therapies; and, 3-months of bilingual outpatient care navigation. Attention control parents receive one in person-education session, monthly well-child texts and usual institutional follow up care. Primary outcome is treatment adherence at 6 months post-discharge measured by percentage of follow-up appointments attended during the prescribed time at hospitals, and community care facilities. Secondary outcomes are functional status of the child using PROMIS parental report measures; and parental health literacy, self-efficacy, and mental health at 3, 6, and 12 months after discharge. Child's academic performance will be assessed using school records. The study evaluates a flexible and scalable intervention using mobile phones to aid transitions of care, improve treatment adherence and TBI outcomes. It addresses the needs of an understudied population and can serve as a model for TBI family centered care for at risk groups.

DETAILED DESCRIPTION:
TBI is a major cause of acquired disability in children. Approximately 60% of children with moderate to severe TBI have long-term cognitive, emotional, or physical deficits. Compared to non-Hispanic children, Hispanic children have higher disability 3 years after TBI, even though differences are not present at hospital discharge. Known risk factors for poor TBI outcomes in children such as underinsurance, low socioeconomic status, and limited parental education are highly prevalent among Hispanics, especially among immigrants from Central America and Mexico. Barriers for receipt of outpatient rehabilitation for Hispanic children are multiple including gaps in understanding of TBI and treatments, limited availability of culturally and linguistically relevant educational resources; and barriers to access services due to transportation, and under-insurance.

Education and navigation programs are efficacious in improving adherence to treatment for children with chronic conditions but have not been tested in children with TBI, despite the need for long-term outpatient rehabilitation. The investigators developed and pilot tested the 1st intervention designed for Hispanic children with TBIs and their families consisting of Brain Injury Education and outpatient Navigation (1st BIEN). The 1st BIEN intervention proposes the novel use of telephone based, culturally relevant patient navigation and education for Hispanic parents of children with TBI. It aims to improve access and adherence to treatment to decrease disability in this high-risk and understudied population. In the 1st BIEN pilot, the investigators established feasibility and acceptability for the program. Now the investigators propose a multicenter randomized controlled trial to test the efficacy of 1st BIEN to maintain long-term adherence to rehabilitation and determine its effect on child's functional outcomes.

Specific aims:

Aim 1. Test the efficacy of the 1st BIEN intervention to improve receipt of overall 1 year follow-up care and outpatient rehabilitation after a TBI among children and adolescents of Hispanic families.

Hypothesis 1a. Intervention group children will have higher attendance at follow-up appointments and higher initiation and attendance at outpatient therapies 6 months after discharge, compared to control children.

Aim 2. Determine the effect of the 1st BIEN intervention on functional outcomes and social participation at 3, 6 and 12 months after TBI hospital discharge among children and adolescents of Hispanic families.

Hypothesis 2a. Intervention group children will have higher adaptive functioning, health related quality of life, better physical, and emotional function, at 3, 6 and 12 months after hospital discharge, compared to control children.

Hypothesis 2b. Intervention group children will have higher levels of social participation measured by earlier school reintegration, receipt of educational resources, and participation in extracurricular activities.

Exploratory Aim 3. Test possible moderators and mediators of 1st BIEN intervention effects. Exploratory analyses will test possible moderators of intervention effects (i.e. pre-injury parental acculturation and education) and possible mediators (i.e. post-intervention parental knowledge, self-efficacy, mental health).

Study design:

Multi-center randomized control trial, enrolling 150 parent-child dyads; Hispanic children 3-17 years of age, hospitalized with a mild, moderate or severe TBI and their primary caregiver parent from 5 centers in Washington, Texas, Dallas, Utah and Oregon. All parents will receive in person education and linguistically and culturally tailored written TBI materials. Intervention parents additionally receive 3 months of Patient Navigation (PN) to support transitions of care and video education through mobile phone devices to promote TBI advocacy skills and reinforce essential TBI knowledge. Control group parents will receive well-child texts once a month to control for attention and follow up per institutional standard of care. Control parents do not receive patient navigation or video education.

Randomization will be done in a 1:1 ratio at each participating institution using a computer-generated random assignment sequence prepared by the study biostatistician and stratified by injury severity (mild complicated; moderate-severe) and age (3-5; 6-11;12-17).

While education using the 1stBIEN booklet is not part of the current usual care at participating institutions, providing all families with initial education at the time of discharge addresses ethical and practical considerations. It standardizes discharge processes at participating institutions while delineating differences in the intensity of education and care coordination activities. The written information given to the attention control group does not equal the amount (dosage) given to the intervention group but provides consistent information to all participants.

Considering that acute processes of care can influence outpatient adherence to treatment and patient outcomes, the investigators will measure institutional and patient level quality indicators of acute rehabilitation care. At the individual level the investigators will measure receipt of inpatient physical, occupational, and speech therapy evaluations and rehabilitation consults; and indicators of family centered care such as assistance with identified needs, telephone counseling services and provision of a contact person for questions after discharge.

Reliability of the intervention will be ensured through meticulous in-person training prior to intervention implementation and monitoring of strict adherence to elements of the intervention. Education of PNs follows a pre-determined curriculum that includes screening and recruitment procedures, inform consent procedures, education of parents using the written materials and using lay language. Training on how to conduct baseline evaluations, scales and forms. After the training PNs should demonstrate proficiency in all procedures, in two case scenarios including use of problem-solving skills during follow-up patient navigation calls, delivery of initial education and delivery of individualized video content education. These tasks will also be monitored on a regular basis via weekly conference calls and complemented by site visits once a year. the investigators will audit twenty percent of PN calls to check for protocol adherence using a standardized checklist. the investigators will audit calls during the first month of implementation of the intervention and then randomly over the 2-year period, following adherence checklists.

ELIGIBILITY:
Children Inclusion criteria:

1. Children 3 to 17 years of age,
2. Hispanic ethnicity
3. Diagnosis of mild, moderate or severe TBI.
4. Hospitalization at one of the 5 academic institutions participating in this trial,
5. Treatment requiring at least one type of rehabilitation therapy as outpatient

Parent Inclusion Criteria:

1. Hispanic ethnicity
2. Being the primary caregiver for the child (For longitudinal follow-up purposes)

Exclusion criteria:

Child:

1. Prior neurological deficits,
2. Acquired brain injuries secondary to other conditions different from trauma.
3. Traumatic brain injuries secondary to abusive trauma.

Parent:

1. Loss of custody of the child (i.e. abusive head trauma)
2. Inability to be contacted by phone

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2022-07-07 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Receipt of follow-up care in centralized Hospital and community | 6 months after discharge.
  Percentage of attended appointments at hospital, primary care and therapies
Child's Health Related Quality of Life | 1 month before injury, 24 hours before discharge from the hospital and 3,6, and 12 months after hospital discharge.
  Pediatric Quality of Life Inventory-PedsQL. A 23-item questionnaire extensively used in TBI outcomes studies. It assesses physical, emotional, social and school functioning. Items on the PedsQL are reverse scored and transformed to a 0-100 scale. Higher scores indicate better health related quality of life, a clinically meaningful difference is 4.5 points. Minimum score is 0 maximum score is 100.

SECONDARY OUTCOMES:
Child's Functional Independence | 24 hours before hospital discharge and through study completion an average of 6 months
  Functional independence measures (FIM) FIM (8+ years) and WeeFIM (3-7 years);18 items (mobility 5 items, self-care 8 items and cognition 5 items) objective functional measures of independence. Every item is scored from"1" (dependent) to "7" (independent).The possible total score ranges from 18 (lowest) to 126 (highest) level of independence. For each item Scores of 1 (total assistance) and 2 (maximal assistance) belong to the "Complete Dependence" category. Scores of 3 (moderate assistance), 4 (minimal contact assistance), and 5 (supervision or set-up) belong to the "Modified Dependence" category. Scores of 6 (modified independence) and 7 (complete independence) belong to the "Independent" category.
Child's Communication | 1 month before injury, 24 hours before discharge from the hospital and 3,6, and 12 months after hospital discharge.
  Adaptive Behavior Assessment System Third Edition (ABAS 3) -Communication subscale. A norm referenced measurement designed to assess adaptive skills. For both subscales, the mean and standard deviation values for healthy individuals are 10 mean and 3SD; higher scores indicate better functioning, and lower scores ,indicate below-average functioning.
Child's Social Skills | 1 month before injury, 24 hours before discharge from the hospital and 3,6, and 12 months after hospital discharge.
  Patient-Reported Outcomes Measurement Information System (PROMIS) Parent Proxy-Peer Relationships (SF7a).Symptoms are rated on a 5-point scale and converted to standard scores. The general population mean is 50 SD 10. Higher scores denote better outcomes.
Child's Anxiety symptoms | 1 month before injury, 24 hours before discharge from the hospital and 3,6, and 12 months after hospital discharge.
  Patient-Reported Outcomes Measurement Information System (PROMIS) Parent Proxy-Anxiety (SF8a) symptoms. Short version of PROMIS parental report pediatric measures of anxiety (8 items). Symptoms are rated on a 5-point scale and converted to standard scores. The general population mean is 50 SD 10. Higher scores denote better outcomes.
Child's Pain Interference | 1 month before injury, 24 hours before discharge from the hospital and 3,6, and 12 months after hospital discharge.
  Patient-Reported Outcomes Measurement Information System PROMIS Parent Proxy-Pain Interference (SF8a). pain interference (8 items).Symptoms are rated on a 5-point scale and converted to standard scores. The general population mean is 50 SD 10. Higher scores denote better outcomes.
Child's Physical Function-Upper Extremity | 1 month before injury, 24 hours before discharge from the hospital and 3,6, and 12 months after hospital discharge.
  Patient-Reported Outcomes Measurement Information System PROMIS Parent Proxy-Physical Function of Upper Extremity (SF8a) .Symptoms are rated on a 5-point scale and converted to standard scores. The general population mean is 50 SD 10. Higher scores denote better outcomes.
Child's Academic Performance | 1 Year before the injury and 1 year after the injury
  School GPA
Child's Fatigue | 1 month before injury, 24 hours before discharge from the hospital and 3,6, and 12 months after hospital discharge
  Patient-Reported Outcomes Measurement Information System PROMIS Parent Proxy - Fatigue (SF 10a). Symptoms are rated on a 5-point scale and converted to standard scores. The general population mean is 50 SD 10. Higher scores denote better outcomes.
Child's Self-care Skills | 1 month before injury, 24 hours before discharge from the hospital and 3,6, and 12 months after hospital discharge.
  Adaptive Behavior Assessment System Third Edition (ABAS 3) - Self-Care subscale. A norm referenced measurement designed to assess adaptive skills. The mean and standard deviation values for healthy individuals are 10 mean and 3SD; higher scores indicate better functioning, and lower scores ,indicate below-average functioning.
Child's Depressive Symptoms | 1 month before injury, 24 hours before discharge from the hospital and 3,6, and 12 months after hospital discharge.
  Patient-Reported Outcomes Measurement Information System (PROMIS) Parent Proxy-Depressive Symptoms (SF6a). Short versions of PROMIS parental report pediatric measures of depression (6 items). Symptoms are rated on a 5-point scale and converted to standard scores. The general population mean is 50 SD 10. Higher scores denote better outcomes.
Child's Mobility | 1 month before injury, 24 hours before discharge from the hospital and 3,6, and 12 months after hospital discharge.
  Patient-Reported Outcomes Measurement Information System PROMIS Parent Proxy-Mobility v2.0 (SF8a).Symptoms are rated on a 5-point scale and converted to standard scores. The general population mean is 50 SD 10. Higher scores denote better outcomes.
Receipt of School support programs | 1 Year before the injury and 1 year after the injury
  School records include information on provision of Individualized Education Programs (IEP), and 504 accommodation plans.

OTHER OUTCOMES:
Parent's Anxiety symptoms | 24 hours before discharge from the hospital and 3,6, and 12 months after hospital discharge.
  Patient-Reported Outcomes Measurement Information System PROMIS Anxiety (SF8b).Symptoms are rated on a 5-point scale and converted to standard scores. The general population mean is 50 SD 10. Higher scores denote better outcomes.
Caregiver Self efficacy | 24 hours before discharge from the hospital and 3,6, and 12 months after hospital discharge.
  The Caregiver Self efficacy (CSE) scale. 7 items scale that measures caregivers' confidence in caring and advocating for patients with brain injuries.
Navigation evaluation | 12 months after discharge from the hospital
  Family Experiences with Coordination of Care (FECC) measurement. A 20-item list of quality indicators of care coordination and engagement with patient navigators for children with medical complexity.
Engagement with video education materials | ongoing tracking (from enrollment - 12 months follow-up)
  Google-analytics
McMaster Family Assessment Device (FAD) | 1 month before injury, 24 hours before discharge from the hospital and 3,6, and 12 months after hospital discharge
  Family general functioning. A 12-item scale that evaluates communication, roles, affective response, involvement and problem solving among families.
Parent's Depressive symptoms | 1 month before injury, 24 hours before discharge from the hospital and 3,6, and 12 months after hospital discharge.
  Patient-Reported Outcomes Measurement Information System PROMIS Depressive Symptoms (SF6b). Symptoms are rated on a 5-point scale and converted to standard scores. The general population mean is 50 SD 10. Higher scores denote better outcomes.
Caregiver Community Self Efficacy (COMSE) | 24 hours before discharge from the hospital and 3,6, and 12 months after hospital discharge.
  Caregiver Community Self-Efficacy (COMSE) measures caregivers' confidence in accessing community services for patients with brain injuries.

CONTACTS AND LOCATIONS:
Overall Officials: Nathalia Jimenez, MD, MPH, Principal Investigator — Seattle Children's Hospital
Locations (6):
- United States (6):
  - Children's Hospital Colorado, Colorado Springs, Colorado
  - Oregon Health & Science University, Portland, Oregon
  - UT Southwestern Medical Center, Dallas, Texas
  - University of Utah, Salt Lake City, Utah
  - Harborview Medical Center - University of Washington, Seattle, Washington
  - Seattle Children's Hospital, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
The 1st BIEN collaborative research group understands and agrees to comply with the NIH policy on Sharing Research Data. The PI and co-investigators from Seattle Children's Research Institute, University of Texas Southwestern Medical Center, Oregon Health and Science University, University of Washington and University of Utah; acknowledge their willingness to share de-identified data from this grant upon request to outside researchers. The database will be produced and will be completely de-identified in accordance with the definitions provided in the Health Insurance Portability and Accountability Act. The Data coordinating center at Seattle Children's will also prepare a data dictionary that provides a brief definition of every data element in the database so that individual investigators will be able to effectively use the data. After approval of 1stBIEN collaborative investigators, IRB and funding agency, controlled access to data will be granted following a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After last subject enrollment and all follow up procedures have been completed, the 1stBIEN collaborative data coordinating center at the Seattle Children's Research Institute will prepare a final study database for the trial, which will then be used for statistical analyses and publication of findings from the trial.
  Our preliminary plan is to release the de-identified underlying primary database at the time of publication of the primary manuscript.
Access Criteria: Access to the releasable database will be in accordance with procedures and regulations of the NIH policy on Sharing Research Data. Release of data will be reviewed by the 1stBIEN collaborative and determined by the scientific merit of the proposal; feasibility, scientific rationale, qualifications and analysis plan; data security protections, and IRB oversight.

REFERENCES:
- [Background] Jimenez N, Fuentes M, Virtue A, Alonso-Gonzalez L, Lopez E, Zhou C, Crawley D, Apkon S, Johnston B, Rivara F. Feasibility and Acceptability of a Telephone-Based Intervention for Hispanic Children to Promote Treatment Adherence After Traumatic Brain Injury: A Pilot Study. J Head Trauma Rehabil. 2021 Jul-Aug 01;36(4):274-281. doi: 10.1097/HTR.0000000000000658. PMID 33656480
- [Derived] Lalji R, Koh L, Francis A, Khalid R, Guha C, Johnson DW, Wong G. Patient navigator programmes for children and adolescents with chronic diseases. Cochrane Database Syst Rev. 2024 Oct 9;10(10):CD014688. doi: 10.1002/14651858.CD014688.pub2. PMID 39382077
- [Derived] Jimenez N, Williams CN, Keenan H, Rinaldi R, Fuentes M, Woodward D, Rivara FP, Zhou C, Ko LK, Bell K. Bilingual randomized controlled trial design, of a telephone-based intervention to promote rehabilitation adherence; A study focus on recruitment of Hispanic children with traumatic brain injury. Contemp Clin Trials. 2023 Dec;135:107362. doi: 10.1016/j.cct.2023.107362. Epub 2023 Oct 16. PMID 37852531